CLINICAL TRIAL: NCT01033981
Title: Cost Effectiveness Of Sunitinib Vs IFN-Alfa Or Bevacizumab + IFN-Alfa As First-Line Treatment In MRCC In Central America And The Caribbean
Brief Title: Cost Effectiveness Of Sunitinib In Central America And Caribbean
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181189
Record Dates: First submitted 2009-12-14; First posted 2009-12-17 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: cost effectiveness; Sunitinib Central America and Caribbean Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Central America and Caribbean: Dominican Republic, Guatemala, Panama, Costa Rica, Honduras, Trinidad & Tobago
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Treatment for mRCC as indication approved and physician criterium

SUMMARY:
Primary Hypothesis: The therapy with Sunitinib represents better cost-effectiveness than IFN-α in first-line treatment for metastatic Renal Cell Carcinoma (mRCC) in Central America and Caribbean countries

DETAILED DESCRIPTION:
This study was terminated on 03Feb2011 due to the fact that the anticipated number of patients expected was not reached. The date of cessation of the drug was January 27, 2011. There was no intervention in the treatment or administration of the drug; the study only observed the treatment and collected data. As the study was dependent on the arrival of new patients with metastatic renal cancer, which was of a very low incidence, the study was terminated. Efficacy, adverse events or other safety issues were not factors in terminating the study. Lack of patients was the only reason.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed (or legally acceptable representative) and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Adult (18 years old or older) men and women with confirmed diagnosis of mRCC treated with Sutent, IFN-α or Bevacizumab + IFN ; on the selected institutions.

Exclusion Criteria:

* Adult men or women with RCCm treated with any other medication that is not Sutent, IFN-α or Bevacizumab + IFN.
* Adult men or women with mRCC with palliative care.
* Adult men or women with RCC without metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and women with mRCC will be evaluated for entering the study. The decision to use Sunitinib, IFN-α or Bevacizumab + IFN must be a joint decision made by the subject and the investigator. The investigator must discuss product information with the subject as per usual practice.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Rate of patients that present metastasis when consulting for first time | 9 months
Rate of use of Sutent, IFN-α and Bevacizumab + IFN-α as first-line treatment | 9 months
Hospitalization average with Sutent, with IFN-α, and with Bevacizumab + IFN-α | 9 months
Rate of success in first-line treatment with Sutent, in first-line treatment with IFN-α and in first-line treatment with Bevacizumab + IFN-α | 9 months
Average number of cycles of Sutent, IFN-α and Bevacizumab + IFN in first-line treatment | 9 months

SECONDARY OUTCOMES:
Percentage of adverse effects with the use of Sunitinib, IFN-α and Bevacizumab + IFN | 9 months
Quality of life in patients using an approved quality questionnaire | 9 months
Costs-benefit of each treatment | 9 months
PFY (progression free years) with each treatment | 9 months
LY (life years) with each treatment | 9 months
QALYs (quality adjusted life years) with each treatment | 9 months
ICER (incremental cost effectiveness ratio) of PFY and LY with each treatment | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Panama City, Panama City, Panama

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181189&StudyName=Cost%20Effectiveness%20Of%20Sunitinib%20In%20Central%20America%20And%20Caribbean